CLINICAL TRIAL: NCT03259607
Title: A Single Dose, Randomized, Four Period, Fasting, Crossover Study to Assess Bioequivalence Between an Oral Nicotine Replacement Product and Nicorette® Mint Gum 2 and 4 mg - in Adult Healthy Male and Female Smokers
Brief Title: Clinical Study to Assess Bioequivalence Between Nicorette Extra Mint Gum and Nicorette® Mint Gum in Healthy Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Collaborators: Janssen (China) Research & Development Center (Unknown)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CO-160307090208-SCCT; 10258820NIK1001 (Other: Janssen TMS)
Record Dates: First submitted 2017-08-02; First posted 2017-08-23 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Tobacco Dependence
Keywords: Bioequivalence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: single-center, randomized, single-dose, open-label, cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): Nicorette Extra Mint 2 mg Gum
  Interventions: Drug: Nicorette Extra Mint 2 mg Gum
- Treatment B (Active Comparator): Nicorette Mint 2 mg Gum
  Interventions: Drug: Nicorette Mint 2 mg Gum
- Treatment C (Experimental): Nicorette Extra Mint 4 mg Gum
  Interventions: Drug: Nicorette Extra Mint 4mg Gum
- Treatment D (Active Comparator): Nicorette Mint 4 mg Gum
  Interventions: Drug: Nicorette Mint 4 mg Gum

INTERVENTIONS:
Drug: Nicorette Extra Mint 2 mg Gum — A single dose of one nicotine gum will be placed on the tongue to be chewed every 2 seconds for 30 minutes.
  Arms: Treatment A
Drug: Nicorette Mint 2 mg Gum — A single dose of one nicotine gum will be placed on the tongue to be chewed every 2 seconds for 30 minutes.
  Arms: Treatment B
Drug: Nicorette Extra Mint 4mg Gum — A single dose of one nicotine gum will be placed on the tongue to be chewed every 2 seconds for 30 minutes.
  Arms: Treatment C
Drug: Nicorette Mint 4 mg Gum — A single dose of one nicotine gum will be placed on the tongue to be chewed every 2 seconds for 30 minutes.
  Arms: Treatment D

SUMMARY:
This is a research study to verify the same effectiveness and safety profile for the test products, nicotine 2 mg gum and nicotine 4 mg gum, as for the already approved products, Nicorette Mint 2 mg gum and Nicorette Mint 4 mg gum (reference products), in a standardized mode. This verification is done in a so-called bioequivalence study, which means that the same amount of the same active substance (nicotine), in the same dosage form, for the same route of administration, and meeting the same or comparable standards is performed.

During the study visits, blood samples will be drawn to measure the level of the substance in the blood to verify that the two test products are comparable to the reference products.

Tolerability of the treatments will be evaluated based on reported and observed adverse events.

DETAILED DESCRIPTION:
This is a single-center, randomized, single-dose open-label, cross-over study in 76 healthy males and females in total. The investigational products (IPs), i.e., Nicorette Extra Mint Gum 2 and 4 mg, and Nicorette Mint Gum 2 and 4 mg, will be given as single doses at separate treatment visits. Investigational treatments will be separated by at least 36 hours.

Blood samples for determination of nicotine will be drawn pre-dose (within 5 minutes of administering, i.e., start of chewing) and at 5, 10, 15, 20, 30, 45, and 60 minutes, as well as 1.5, 2, 4, 6, 7, 8, 9, and 10 hours after start of administration.

Used gums will be collected and analyzed to determine the amount of remaining nicotine.

Any Adverse Events (AEs) that may occur will be registered.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 18 and 55 years, inclusive, and healthy female subjects between the ages of 18 and 45 years, inclusive. Health is defined as the absence of clinically relevant abnormalities identified by a detailed medical history, physical examination, blood pressure and pulse rate measurements, 12-lead electrocardiogram (ECG) as well as clinical laboratory tests, as judged by the Investigator or an authorized physician.
2. Smoking of at least 10 cigarettes daily for at least one year preceding inclusion.
3. Subjects will have a body mass index (BMI) between 19 and 25 (inclusive) kg/m2 and a body weight >50 kg.
4. Females of childbearing potential must have a negative pregnancy test at the screening visit.
5. Male or non-pregnant, non-lactating female agree to the contraceptive requirements including male's and female partner's use of a highly effective methods of birth control for at least 3 months before the study, during the study and for 30 days after the last dose of the study drug).
6. A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study before participating in any study-specific procedures.
7. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures specified in the protocol.

Exclusion Criteria:

1. Use of medications other than contraceptives specified in Inclusion Criterion 4. Vitamins, dietary, and herbal supplements must be discontinued at least two days before the first dose of study medication.
2. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, Human Immunodeficiency Virus (HIV) or syphilis.
3. Hypersensitivity to the ingredients/components of any of the IPs.
4. History of alcoholism, as judged by the Investigator, within the past 6 months preceding this study and/or presenting a positive respiratory alcohol test (breathalyzer) at the screening visit.
5. History of drug abuse or presenting a positive drug screening test for psychoactive drugs and narcotic substances at screening visit.
6. Treatment with an IP within 3 months preceding this study.
7. Donation or loss of blood within 3 months preceding this study if the estimated lost blood volume equaled or exceeded 200 mL.
8. Impaired chewing capability as assessed by oral examination (e.g. dentures, significant oral ulceration) or impaired salivary secretion (e.g. Sicca syndrome). Piercing of tongue and lips is considered to impair oral function.
9. Preplanned surgery or procedures during the study period, if this may interfere with the conduct of the study.
10. Relationship to persons involved directly with the conduct of the study (i.e. PI; Sub investigators; study coordinators; other study personnel; employees or contractors of the sponsor or Johnson & Johnson (J&J) subsidiaries; and the families of each).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of nicotine. | At baseline, 5, 10, 15, 20, 30, 45, and 60 minutes, as well as 1.5, 2, 4, 6, 7, 8, 9, and 10 hours after start of administration.
  The maximum observed plasma concentration (Cmax).
Area under the plasma concentration versus time curve (AUCt) from start of nicotine administration until the last measurable concentration. | At baseline, 5, 10, 15, 20, 30, 45, and 60 minutes, as well as 1.5, 2, 4, 6, 7, 8, 9, and 10 hours after start of administration.
  AUCt is defined as area under the plasma concentration versus time curves from start of drug administration until the last measureable concentration.
Area under the plasma concentration versus time curve (AUC∞) of nicotine. | At baseline, 5, 10, 15, 20, 30, 45, and 60 minutes, as well as 1.5, 2, 4, 6, 7, 8, 9, and 10 hours after start of administration.
  AUC∞ is defined as area under the plasma concentration versus time curves from start of drug administration until the nicotine plasma concentration is negligible (infinity).

SECONDARY OUTCOMES:
The extrapolated part of area under the plasma concentration versus time curve (AUC∞) of nicotine. | Extrapolation from 12 hours after start of drug administration until 48 hours.
  The area under the plasma concentration versus time curves from start of drug administration until 48 hours (infinity).
The time at which the maximum nicotine concentration (Cmax) occurs (Tmax). | At baseline, 5, 10, 15, 20, 30, 45, and 60 minutes, as well as 1.5, 2, 4, 6, 7, 8, 9, and 10 hours after start of administration.
  Tmax is defined as the time point at which the maximum nicotine concentration (Cmax) occurs.
Determination of the terminal elimination rate constant (lambda_z) for nicotine. | At baseline, 5, 10, 15, 20, 30, 45, and 60 minutes, as well as 1.5, 2, 4, 6, 7, 8, 9, and 10 hours after start of administration.
  The rate at which the drug is removed from the body system.
The plasma half-life (t1/2) of nicotine. | At baseline, 5, 10, 15, 20, 30, 45, and 60 minutes, as well as 1.5, 2, 4, 6, 7, 8, 9, and 10 hours after start of administration.
  The time taken for the nicotine plasma concentration to fall to half its original value.
Amount of nicotine extracted from Nicorette Mint 2 mg gums. | After 30 minutes of chewing.
  The residual amount of nicotine in the chewed gums will be analyzed and subtracted from the original amount of nicotine in the gums, and summarized descriptively.
Amount of nicotine extracted from Nicorette Mint 4 mg gums. | After 30 minutes of chewing.
  The residual amount of nicotine in the chewed gums will be analyzed and subtracted from the original amount of nicotine in the gums, and summarized descriptively.
Amount of nicotine extracted from Nicorette Extra Mint 2 mg gums. | After 30 minutes of chewing.
  The residual amount of nicotine in the chewed gums will be analyzed and subtracted from the original amount of nicotine in the gums, and summarized descriptively.
Amount of nicotine extracted from Nicorette Extra Mint 4 mg gums. | After 30 minutes of chewing.
  The residual amount of nicotine in the chewed gums will be analyzed and subtracted from the original amount of nicotine in the gums, and summarized descriptively.
Percentage of Subjects with Treatment-Emergent Adverse Events after single-dose administration of investigational product. | From first dose received up to 2.5 weeks + 30 days follow up after study completion for any unresolved adverse events.
  Percentage of subjects experiencing treatment-emergent adverse events by treatment, system organ class and preferred term.
Percentage of Subjects with Treatment-Emergent Adverse Events after single-dose administration of investigational product - by worst-case severity. | From first dose received up to 2.5 weeks + 30 days follow up after study completion for any unresolved adverse events.
  Percentage (%) of subjects experiencing treatment-emergent adverse events by treatment, system organ class, preferred term and severity.
Percentage of Subjects with common treatment-emergent adverse events (AEs) after single-dose administration of Investigational product. | From first dose received up to 2.5 weeks + 30 days follow up after study completion for any unresolved adverse events.
  Percentage (%) of subjects with commonly reported treatment-emergent adverse events by system organ class and preferred term.
Percentage of Subjects with treatment-related adverse events (AEs) after single-dose administration of investigational product. | From first dose received up to 2.5 weeks + 30 days follow up after study completion for any unresolved adverse event.
  Percentage (%) of subjects experiencing treatment-related adverse events by treatment, system organ class and preferred term.
Percentage of Subjects with treatment-related adverse events (AEs) after single-dose administration of investigational product - by worst-case severity. | From first dose received up to 2.5 weeks + 30 days follow up after study completion for any unresolved adverse events.
  Percentage (%) of subjects experiencing treatment-related adverse events by treatment, system organ class, preferred term and severity.
Percentage of Subjects with treatment-emergent serious adverse events (SAEs). | From first dose received up to 2.5 weeks + 30 days follow up after study completion.
  Percentage (%) of subjects experiencing treatment-emergent serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Shi Aixin, M. Pharm, Principal Investigator — BeiJing Hospital, No.1, Beijing, China.
Locations (1):
- Beijing Hospital, No.1, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CO-160307090208-SCCT&attachmentIdentifier=c6a9db7d-71aa-4100-9101-9dce03e91cd3&fileName=Polar_Bear_CSR_Synopsis_redacted_CT.GOV_registration_of_Results_Redacted_PDFA.pdf&versionIdentifier=